CLINICAL TRIAL: NCT00442598
Title: An Open-Label Phase 2 Study of the Safety and Efficacy of Glufosfamide in Ovarian Cancer
Brief Title: Safety and Efficacy Study of Glufosfamide in Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Eleison Pharmaceuticals LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-303
Record Dates: First submitted 2007-02-28; First posted 2007-03-02 (Estimated); Results first posted 2015-03-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Ovarian Cancer
Keywords: Ovarian; Cancer; CA-125; Third-line; Glufosfamide
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — beta-D-glucosylisophosphoramide mustard

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glufosfamide q21 days (Experimental): 1-hour infusion of glufosfamide at a dose of 5,000 mg/m2 on Day 1 of a 21-day cycle
  Interventions: Drug: Glufosfamide
- Glufosfamide q7 days low (Experimental): 1-hour infusion of glufosfamide at a dose of 1,660 mg/m2 on Days 1, 8 and 15 of a 21-day cycle
  Interventions: Drug: Glufosfamide
- Glufosfamide q7 days high (Experimental): 1-hour infusion of glufosfamide at a dose of 2,500 mg/m2 on Days 1, 8 and 15 of a 21-day cycle
  Interventions: Drug: Glufosfamide

INTERVENTIONS:
Drug: Glufosfamide

SUMMARY:
Primary Objectives:

* To evaluate the effect of glufosfamide on the serum concentrations of CA125 in subjects with ovarian cancer
* To evaluate the safety of weekly glufosfamide dosing in subjects with ovarian cancer as compared with every 21-day dosing

Secondary objectives:

* To evaluate the efficacy of glufosfamide in subjects with ovarian cancer as measured by objective response rate, duration of response, progression-free survival, and overall survival
* To evaluate the pharmacokinetics of glufosfamide and isophosphoramide mustard during and after treatment

Exploratory objective:

* To correlate efficacy endpoints with expression of tumor-associated glucose transporter proteins

DETAILED DESCRIPTION:
Open-label, multicenter, Phase 2 dose escalation study. Subjects will be randomized to receive either once every three weeks dosing regimen or the weekly dosing regimen. Randomization will utilize a 2:1 ratio with two-thirds of the subjects randomized to the weekly dosing regimen.

In the weekly dosing schedule, treatment with glufosfamide 2,500 mg/m2 will be initiated only after the 1,660 mg/m2 treatment cohort has been enrolled and there is evidence that the dose of 1,660 mg/m2 has been well tolerated (See below Section on Pharmacokinetic/Statistical Analyses).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee
* Pathologically confirmed epithelial ovarian cancer, peritoneal serous cancer, or carcinoma of the fallopian tube
* Prior treatment with at least one platinum-based chemotherapy
* Evidence of resistance to most recent platinum-containing regimen (relapsed during or within 6 months after completing chemotherapy)
* Evidence of CA 125 progression after most recent chemotherapy defined as either:

  * CA 125 at least 40 U/mL for patients with elevated CA 125 that decreased to <20 U/mL on therapy; or
  * CA 125 at least 40 U/mL and at least a 50% increase over the nadir value for patients with elevated CA 125 that did not decrease to <20 U/mL on therapy.

CA 125 must meet criteria on two occasions not less than one week apart if the CA 125 has increased by at least 100% (i.e., doubled). There must be 3 consecutive increasing measurements over a period of at least two weeks if the CA 125 has increased by at least 50% but less than 100%.

* Elevated serum CA125 (≥40 U/mL) within 2 weeks prior to starting treatment
* At least one target or nontarget lesion by RECIST
* A minimum of 21 days between prior chemotherapy, radiation therapy, immunotherapy, or other anti-tumor therapy and study entry
* Recovered from reversible toxicities of prior therapy
* ECOG score of 0 or 1
* ANC ≥ 1,500/µL, platelets ≥ 100,000/µL, hemoglobin ≥9 g/dL
* Total bilirubin ≤ 1.5-fold ULN, AST/ALT ≤ 2.5-fold ULN (≤ 5-fold ULN if liver metastases)
* Creatinine clearance ≥ 60 mL/min (calculated by Cockcroft-Gault formula)
* All women of childbearing potential must have a negative serum pregnancy test and must agree to use effective means of contraception (surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) from entry into the study through 6 months after the last dose

Exclusion Criteria:

* Concomitant or planned hormonal therapy, radiation therapy, biologic therapy, chemotherapy or other systemic antitumor therapy for ovarian cancer other than protocol therapy
* Symptomatic brain metastases
* Active clinically significant infection requiring antibiotics
* Known HIV positive or active hepatitis B or C
* Recent (one year) history or symptoms of cardiovascular disease (NYHA Class 2, 3, or 4), particularly coronary artery disease, arrhythmias or conduction defects with risk of cardiovascular instability, uncontrolled hypertension, clinically significant pericardial effusion, congestive heart failure or stroke
* Other active malignancies (other than treated non-melanoma skin cancer or treated in situ cancer) within the past 5 years
* Major surgery within 3 weeks of the start of study treatment, without complete recovery
* Females who are pregnant or breast-feeding
* Participation in an investigational drug or device study within 28 days of the first day of dosing on this study
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Unwillingness or inability to comply with the study protocol for any other reason

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Alberts, MD, Principal Investigator — University of Arizona; Michael Gordon, MD, Principal Investigator — Premiere Oncology of Arizona; Daniela Matei, MD, Principal Investigator — Indiana University School of Medicine; Peter D Eisenberg, MD, Principal Investigator — California Cancer Center; Larry Puls, MD, Principal Investigator — Gynecologic Oncology Research & Development, LLC; Krishnansu Tewari, MD, Principal Investigator — UCI Chao Family Comprehensive Cancer Center; Nashat Gabrail, MD, Principal Investigator — Gabrail Cancer Center; Jeffrey Goldberg, MD, Principal Investigator — Louisville Oncology Clinical Research Program; Claire Verschraegen, M.D., Principal Investigator — New Mexico Cancer Research Alliance; William Robinson, MD, Principal Investigator — Harrington Cancer Center
Locations (10):
- United States (10):
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - California Cancer Center, Greenbrae, California
  - UCI Chao Family Comprehensive Cancer Center, Orange, California
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Louisville Oncology Clinical Research Program, Louisville, Kentucky
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Gabrail Cancer Center, Canton, Ohio
  - Gynecologic Oncology Research & Development, LLC, Greenville, South Carolina
  - Harrington Cancer Center, Amarillo, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Glufosfamide q21 Days: 1-hour infusion of glufosfamide at a dose of 5,000 mg/m2 on Day 1 of a 21-day cycle
  Glufosfamide
- Glufosfamide q7 Days Low: 1-hour infusion of glufosfamide at a dose of 1,660 mg/m2 on Days 1, 8 and 15 of a 21-day cycle
  Glufosfamide
- Glufosfamide q7 Days High: 1-hour infusion of glufosfamide at a dose of 2,500 mg/m2 on Days 1, 8 and 15 of a 21-day cycle
  Glufosfamide
Period: Overall Study
Arm/Group | Glufosfamide q21 Days | Glufosfamide q7 Days Low | Glufosfamide q7 Days High
Started | 7 | 10 | 0
Two Cycles | 5 | 6 | 0
Completed | 1 | 2 | 0
Not Completed | 6 | 8 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Tumor progression | 3 | 4 | 0
Not completed — Clinical deterioration | 1 | 2 | 0
Not completed — CA125 progression | 0 | 1 | 0
Not completed — Reduced creatinine clearance | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glufosfamide q21 Days | Glufosfamide q7 Days Low | Glufosfamide q7 Days High | Total
Number analyzed (Participants) | 7 | 10 | 0 | 17
Age, Categorical [Number; unit: participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 6 | 6 |  | 12
  >=65 years | 1 | 4 |  | 5
Age, Continuous [Median (Full Range); unit: years] | 60 [44 to 74] | 52 [40 to 67] |  | 58 [40 to 74]
Gender [Number; unit: participants]
  Female | 7 | 10 |  | 17
  Male | 0 | 0 |  | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 0 |  | 0
  White | 7 | 10 |  | 17
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: CA 125 Response Rate
Description: Reduction in blood levels of CA 125 of >50% from baseline, confirmed at the next study cycle.
Time Frame: Duration of study, up to 18 weeks.
Measure: Number; unit: participants
Arm/Group | Glufosfamide q21 Days | Glufosfamide q7 Days Low | Glufosfamide q7 Days High
Number analyzed (Participants) | 7 | 10 | 0
participants
  Partial response | 1 | 0 |
  Stable disease | 6 | 10 |

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate measured by RECIST v1.0
Time Frame: Duration of study, up to 18 weeks.
Measure: Number; unit: participants
Arm/Group | Glufosfamide q21 Days | Glufosfamide q7 Days Low | Glufosfamide q7 Days High
Number analyzed (Participants) | 7 | 10 | 0
participants
  Stable disease | 3 | 3 |
  Progressive disease | 4 | 7 |

3. Secondary Outcome: Progression-free Survival
Description: Time from initiation of study drug to disease progression or death on study
Time Frame: Median measured in months
Measure: Median (Full Range); unit: months
Arm/Group | Glufosfamide q21 Days | Glufosfamide q7 Days Low | Glufosfamide q7 Days High
Number analyzed (Participants) | 7 | 10 | 0
months | 1.2 [0.7 to 4.6] | 1.9 [0.0 to 4.5] |

4. Secondary Outcome: Overall Survival
Description: Time from initiation of study drug to death.
Time Frame: Median measured in months, until death or censorship at analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Glufosfamide q21 Days | Glufosfamide q7 Days Low | Glufosfamide q7 Days High
Number analyzed (Participants) | 7 | 10 | 0
months | 5.6 [1.6 to 13.7] | 6.8 [0.9 to 8.5] |

ADVERSE EVENTS:
Arm/Group | Glufosfamide q21 Days | Glufosfamide q7 Days Low
Serious Adverse Events (participants affected / at risk) | 2/7 | 3/10
Other Adverse Events (participants affected / at risk) | 7/7 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glufosfamide q21 Days (N=7) | Glufosfamide q7 Days Low (N=10)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glufosfamide q21 Days (N=7) | Glufosfamide q7 Days Low (N=10)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Lymphadenitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Tumor associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (6) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Decreased apetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3)
Headache (Nervous system disorders) | 2 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (2)
Visual field defect (Nervous system disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (10) | 4 (5)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (2) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Catheter related complication (General disorders) | 1 (4) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (2) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (8) | 4 (5)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Performance status decreased (General disorders) | 0 (0) | 1 (1)
Temperature intolerance (General disorders) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Feeding tube complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No